CLINICAL TRIAL: NCT03498300
Title: Seroprevalence of Bordetella Pertussis Antibodies and Anti-pertussis Antibody Response After a Single Dose of Reduced-antigen, Combined Diphtheria, Tetanus, and Acellular Pertussis Vaccine (Tdap) in Pregnant Thai Women
Brief Title: Seroprevalence of Bordetella Pertussis Antibodies and Anti-pertussis Antibody Response After a Single Dose of Tdap in Pregnant Thai Women
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Nalat Sompagdee, Principal Investigator, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SI 089/2018
Record Dates: First submitted 2018-04-07; First posted 2018-04-13 (Actual); Results first posted 2020-03-24 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Pertussis; Pregnancy Related
MeSH Terms: conditions — Whooping Cough

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Experimental (Experimental): A single dose of Tdap vaccine at GA 27 - 36 weeks
  Interventions: Biological: Tdap vaccine
- Active comparator (No Intervention): dT vaccine as standard protocol

INTERVENTIONS:
Biological: Tdap vaccine — A single dose of Tdap vaccine at GA 27 - 36 weeks
  Arms: Experimental

SUMMARY:
This study evaluated the seroprevalence of Bordetella pertussis antibodies and anti-pertussis antibody response after a single dose of reduced-antigen, combined diphtheria, tetanus, and acellular pertussis vaccine (Tdap) in pregnant Thai women.

All seronegative participants received Tdap, while seropositive participants were equally randomized into 2 groups. Half of seropositive participants received Tdap and the other half received tetanus-diphtheria (Td) as standard protocol.

DETAILED DESCRIPTION:
The primary objective of this study was to determine the seroprevalence of anti-pertussis toxin antibodies (anti-PT IgG) among pregnant Thai women. The secondary objectives were to evaluate antibody response after Tdap vaccination between seronegative and seropositive participants and to compare the different antibody titers at delivery among seropositive participants who received Tdap to those who received tetanus-diphtheria vaccine (Td). The sample size calculation was based on the primary objective. Randomized clinical trial was performed for the latter secondary objective.

ELIGIBILITY:
Inclusion Criteria:

* Thai pregnant women age at least 18 years
* No known underlying disease
* Singleton pregnancy without maternal or fetal complications
* Gestational age not more than 20 weeks at the time of recruitment
* Desired for delivery at Siriraj Hospital

Exclusion Criteria:

* Pregnant women who have any contraindication to Tdap vaccine including

  1. History of serious allergic reaction to any components of Tdap vaccine
  2. History of seizure or coma after receiving Tdap vaccine in childhood
  3. Having an underlying disease involving central nervous system (e.g., epilepsy, Guillain-Barré syndrome)
* History of serious reactions after receiving Tdap vaccine (e.g., severe pain, severe swelling at the injection site)
* Recently had Tdap vaccine injection
* Denied for Tdap vaccine injection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2018-05-09 (Actual); Primary Completion 2019-04-13 (Actual); Study Completion 2019-04-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nalat Sompagdee, MD, Principal Investigator — Mahidol University
Locations (1):
- Nalat Sompagdee, Bangkok Noi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The sample size of 129 participants was calculated based on the primary objective. Randomized clinical trial on 42 seropositive participants was performed for one of the secondary objectives, which was to compare the different anti-PT IgG at delivery among seropositive participants who received Tdap to those who received Td.
Period: Overall Study
Arm/Group | Experimental | Active Comparator
Started | 21 | 21
Completed | 18 | 13
Not Completed | 3 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental | Active Comparator | Total
Number analyzed (Participants) | 18 | 13 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.8 (7.4) | 28.5 (6) | 29.2 (6.8)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 18 | 13 | 31
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: The Seroprevalence of Anti-pertussis Toxin Antibodies (Anti-PT IgG) in Pregnant Thai Women
Description: Percentage of participants who were seropositive for anti-pertussis toxin antibodies (anti-PT IgG).
  The overall number of 129 participants is greater than the number of 42 participants include in the Particiant Flow Module because it was the sample size calculated based on the primary objective, which was the seroprevalence of anti-pertussis antibodies in pregnant Thai women. Randomized clinical trial on 42 seropositive participants was performed for one of the secondary objectives, which was to compare the different anti-PT IgG at delivery among seropositive participants who received Tdap to those who received Td.
Time Frame: Four months
Measure: Count of Participants; unit: Participants
Groups:
- All Participants: After enrollment, a blood sample was obtained for determination of anti-PT IgG on the day of the first antenatal visit from all of the participants. If the anti-PT IgG level was 5 international units per milliliter (IU/ml) or more, the woman was considered to have seropositivity.
Arm/Group | All Participants
Number analyzed (Participants) | 129
Participants | 43

2. Secondary Outcome: Change From Baseline in Anti-pertussis Toxin Immunoglobulin G Levels Among Seropositive Participants Who Received Tdap to Those Who Received Td
Time Frame: Eight months
Measure: Median (Inter-Quartile Range); unit: IU/ml
Arm/Group | Experimental | Active Comparator
Number analyzed (Participants) | 18 | 13
IU/ml | 42 [16.7 to 65.2] | -7.4 [-14.3 to -6.3]

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 11 months
Arm/Group | Experimental | Active Comparator
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/13
Other Adverse Events (participants affected / at risk) | 12/18 | 12/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental (N=18) | Active Comparator (N=13)
Gestational diabetes (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 3 (3)
Preterm delivery (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0)
Threatened preterm labor resulting in hospitalization (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 1 (1)
Postpartum hemorrhage (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Congenital defects (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 2 (2)
1-minute Apgar score of 7 or less (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 1 (1)
Prolonged hospitalization of the newborn after birth (more than 7 days) (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-11): https://cdn.clinicaltrials.gov/large-docs/00/NCT03498300/Prot_SAP_000.pdf